CLINICAL TRIAL: NCT02134041
Title: Observational Study for Amyloid Accumulation After Mild Traumatic Brain
Brief Title: Amyloid Accumulation After Mild Traumatic Brain Injury
Acronym: TBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chaur-jong Hu, Chief, Department of Neurology, Taipei Medical University Shuang Ho Hospital
Other Study IDs: DOH101-TD-PB-111-NSC017; DOH101-TD-PB-111-NSC017 (Other Grant/Funding Number: National Scince council of Taiwan)
Record Dates: First submitted 2012-10-15; First posted 2014-05-08 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Traumatic Brain Injury; Dementia; Alzheimer Disease
Keywords: traumatic brain injury; Alzheimer disease
MeSH Terms: conditions — Brain Injuries, Traumatic; Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — peripheral blood for APOE genotyping
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- traumatic brain injury: mild traumatic brain injury
  Interventions: Other: traumatic brain injury
- without TBI: without TBI

INTERVENTIONS:
Other: traumatic brain injury — mild TBI, GCS >/=13 after traumatic brain injury
  Other Names: TBI
  Groups: traumatic brain injury

SUMMARY:
We are extending the researches of Taiwan neurosurgery traumatic brain injury (TBI) database which is led by Professor WT Chiu in Taipei Medical University and will recruit mild TBI (mTBI) participants who have ever been registered in the database. This database has been established for over 15 years and contains the information of over 150000 patients. It is one of the largest TBI database in the world.

TBI usually results from traffic accidents, falls or violence events. Most of the victims are young people and the victims suffer from life-threatening and mental-physical deficits. Mild TBI (mTBI) usually was neglected before because its symptoms, signs are mild and mTBI patients usually were not obtained enough initial treatment. Therefore, mTBI might result in long-term cognitive and affective impairments, such as depression, indifference, anxiety, memory impairment, loss of attention and executive function. These late effects not only decrease the life quality of patients and their family but also increase the social and medical burden.

Recent epidemiology studies have pointed out that TBI would increase the risk for dementia, especially Alzheimer disease (AD) by 2-4 times. However, the association between TBI severity, number of repeats, genetic factors and onset of AD remains further investigation.

Amyloid-β (Aβ) plaques and neurofibrillary tangles are the pathological hallmarks for AD. Accumulation of Aβ is considered to be the first step of pathophysilogy of AD. Compelling researches have supported TBI accelerates the formation and accumulation of Aβ. These findings could link TBI with AD but the previous researches had limitations. There was lack of mTBI pathology data so the impacts of mTBI on Aβ accumulation were still obscure. By amyloid-PET, we could study the effects of mTBI on the accumulation of Aβ and this tool could be helpful for understanding the real impacts and pathophysiological mechanisms of mTBI on AD.

DETAILED DESCRIPTION:
We will conduct amyloid PET, cognitive examination and APOE genotyping for the individuals who had traumatic brain injury (TBI) in 1 year, 5 years, 10 years and 15 years ago. Age-gender-matched controls without TBI will be recruited.

The main aim of this study is to evaluate the impact of TBI on amyloid accumulation in the brain. In the mean time, we also will test the effects of APOE genotypes in amyloid accumulation after TBI and the clinical relevants, in terms of cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* a. had TBI in 1, 5, 10 and 15 years ago b. mild injury in TBI (initial GCS = 13-15) c. had MRI or CT evaluation after TBI d. aged 18 years or older (55 years better) e. have agreement and have signed the informed consent form by him/herself or his/her legal representative

Exclusion Criteria:

* a. participating in another clinical trials which might interfere the current finding b. not sure the timing of TBI c. contaminant the symptoms with injury, skull fracture, intracranial hemorrhage, craniotomy, and death d. moderate (initial GCS = 9-12) or severe (initial GCS < 8) injury in TBI e. had wound with gunshot or puncture f. loss of consciousness over 30 minutes after TBI g. loss of memory for over 1 day after TBI h. have no MRI or CT evaluation of brain after TBI or have obstructive ischemia after MRI or CT evaluation i. have uremia, liver cirrhosis, heart failure, pulmonary edema, coagulation disorders and other major diseases j. pregnant woman or emotional instability k. the age less than 18 years (55 years better) l. unable to collect blood sample by peripheral vein m. determination of inappropriate participants in the clinical trail of PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients aged over 55 years with/without traumatic brain injury 1, 5, 10, 15 years ago
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-10; Primary Completion 2019-08 (Actual); Study Completion 2019-09-18 (Estimated)

PRIMARY OUTCOMES:
amyloid accumulation by amyloid PET | day one
  amyloid PET after participation

SECONDARY OUTCOMES:
mini-mental status examination (MMSE) for cognitive function | day one
  neuro-psychological test by use of mini-mental status examination (MMSE) to measure the cognitive function of participants

OTHER OUTCOMES:
APOE genotypes | day one

CONTACTS AND LOCATIONS:
Overall Officials: Chaur-Jong Hu, M.D., Principal Investigator — Department of Neurology, Shuang Ho Hospital, Taipei medical University
Locations (1):
- Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

REFERENCES:
- [Background] Lin KJ, Hsu WC, Hsiao IT, Wey SP, Jin LW, Skovronsky D, Wai YY, Chang HP, Lo CW, Yao CH, Yen TC, Kung MP. Whole-body biodistribution and brain PET imaging with [18F]AV-45, a novel amyloid imaging agent--a pilot study. Nucl Med Biol. 2010 May;37(4):497-508. doi: 10.1016/j.nucmedbio.2010.02.003. Epub 2010 Apr 7. PMID 20447562